CLINICAL TRIAL: NCT04842864
Title: Time Course for Fasting-induced Autophagy in Humans
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: According to the PI/Responsible Party no participants were able to be enrolled into the study following approval.
Sponsor: Montefiore Medical Center (Other)
Collaborators: Glenn Foundation for Medical Research (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2021-12857
Record Dates: First submitted 2021-04-06; First posted 2021-04-13 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Fasting; Autophagy; Aging Well; Ketosis, Metabolic
MeSH Terms: conditions — Fasting; Ketosis | interventions — Angptl4 protein, mouse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Young (Experimental): 10 healthy men and women 18-35 yo.
  Interventions: Behavioral: Fasting
- Older adults (Active Comparator): 10 healthy men and women 65-85 yo
  Interventions: Behavioral: Fasting

INTERVENTIONS:
Behavioral: Fasting — 23 hours fasting

SUMMARY:
Autophagy, which involves the degradation of aged or damaged cellular components, has been shown to extend healthspan and lifespan in multiple organisms, including flies, worms, and mice. Research has also demonstrated that autophagy declines with age in these simpler experimental models. However, human studies are lacking. Our study seeks to determine whether fasting, a robust stimulus of autophagy, upregulates autophagy in humans, and whether autophagy is reduced in healthy older people compared to healthy younger individuals.

DETAILED DESCRIPTION:
Autophagy is a cellular quality control pathway that degrades aged or damaged organelles and protein aggregates within lysosomes. By doing so, autophagy provides an alternate source of energy for cells to cope with adverse conditions. The level of autophagy determines the degree to which aged cells are able to eliminate damaged organelles and/or toxic aggregates and mount a protective response against stress. At the physiological level, nutrient deprivation or fasting is one of the most robust stimuli for autophagy across diverse experimental systems.1 Our lab has shown important roles for autophagy in lipid/glucose homeostasis and regulation of energy balance. We have found that autophagy degrades cellular lipid stores via a process we described as lipophagy. We have also shown contributions of autophagy to the regulation of feeding as well as its developmental roles in maintenance of muscle and fat mass. In addition to these physiological functions, a number of studies have revealed that mice lacking autophagy in the central nervous system show rapid onset of neurodegeneration and an early death.2,3 These studies support a central role of autophagy in the maintenance of healthspan.

It is well-established that autophagy activity declines with age, which has led to the hypothesis that autophagy failure contributes to the metabolic syndrome of aging. In fact, young mice with tissue-specific knockout of the autophagy gene Atg7 display features of aging, including loss of muscle mass (mimicking sarcopenia of aging), fatty liver, decreased adipose lipolysis, de-differentiation of brown fat, and pancreatic β-cell dysfunction.4-6 Conversely, restoration of autophagy via pharmacological or genetic approaches prevents age-associated decline in cell function and improves stress response-thus directly extending healthspan. As a consequence, there is great interest in developing new experimental approaches to prevent age-associated chronic diseases. In fact, caloric restriction (CR) has been shown to stimulate autophagy and extend lifespan and healthspan in multiple experimental models. While these CR studies were carried out in simpler organisms, such as flies, worms, and mice,7-9 similar studies in humans are largely lacking. Since autophagy is activated by starvation, the prevailing hypothesis is that caloric restriction (CR) or more physiological approaches such as intermittent fasting will stimulate autophagy in humans, which in turn will prevent or retard the onset of age-associated chronic diseases. There is limited knowledge if indeed extended periods of fasting will activate autophagy in humans. In addition, we do not know what duration of fasting may be required to stimulate autophagy in humans. Finally, we do not know if, nor by how much, fasting-induced autophagy is reduced in aging humans. Due to the aforementioned gaps in our knowledge regarding autophagy in humans, in this study we will test the ability of extended periods of restriction to food to stimulate autophagy in healthy, young individuals. Further, we will compare the extent to which autophagy is reduced in healthy older subjects, when compared to those observed in young controls. In our study, we will be using samples of adipose tissue, a metabolically active endocrine organ, and peripheral blood cells, which have both been evaluated in prior autophagy studies and can be obtained in a less invasive manner.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women 18-35 years of age
* Healthy men and women 65-85 years of age

Exclusion Criteria:

* Serious acute/chronic illness (e.g., active cancer, inflammatory states, RA, SLE, or a CVD event within past 6 months)
* Diabetes or pre-diabetes with an A1c >6.0%
* Pregnancy
* BMI >30 kg/m2 or <20 kg/m2
* eGFR <45 ml/min
* ALT >3x ULN
* Hct <35 or Hb <10
* Exclusionary meds: calcium channel blockers, anticonvulsants or other drugs shown to affect autophagy (see table below)
* Food allergy or known food intolerance
* Active Smoking (>1 cigarette or cigar per week)
* Use of recreational drugs (opioids, cocaine, marijuana, etc.) in past month
* Use of alcohol on the day prior to and the day of study
* Shift workers or other dysregulated sleep pattern (habitual use of sleep medications, jet lag, etc.)
* Strenuous exercise within 3 days prior to study visit 2
* Any condition the investigator believes would impair the ability to interpret targeted outcomes

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11-19 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Autophagy flux | 23 hours
  The turnover rate of the autophagosome marker LC3-II will be assessed. LC3-II flux will be performed in freshly isolated fat tissues and in PBMCs at various timepoints. Freshly collected fat tissue explants and PBMCs will be incubated in dishes with high-glucose culture medium (DMEM) in the presence or absence of lysosomal inhibitors (Lys Inh), leupeptin (200uM) and ammonium chloride (20uM) at 37°C, 5% CO2 for 4 hours. Fat explants and scraped PMBC pellets will then be homogenized in a buffer containing protease and phosphatase inhibitors and subjected to immunoblotting for LC3. Autophagy flux will be determined by subtracting the densitometric value of LC3-II in Lys Inh-untreated samples from the Lys Inh-treated samples.

SECONDARY OUTCOMES:
Level of ketone bodies | 23 hours
  Levels of ketones in the plasma will be assessed with blood draws at various timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: Jill Crandall, MD, Principal Investigator — Albert Einstein College of Medicine; Nir Barzilai, MD, Principal Investigator — Albert Einstein College of Medicine; Rajat Singh, MD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No